CLINICAL TRIAL: NCT01033136
Title: Exposure Therapy for Veterans With PTSD and Panic Attacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CDA2-012-09F
Record Dates: First submitted 2009-12-03; First posted 2009-12-16 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-08

CONDITIONS: PTSD; Panic Attacks
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Panic Disorder | interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Intervention Model Description: Multiple Channel Exposure Therapy is a behavioral treatment that simultaneously targets panic disorder and PTSD.
Who Masked: Outcomes Assessor
Masking Description: Post-treatment and follow-up assessments are conducted by an assessor masked to treatment condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MCET-V (Experimental): Multiple Channel Exposure Therapy -Veterans (MCET-V) is a 12-session cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks. It is an integrated treatment designed to target panic and PTSD symptoms simultaneously.
  Interventions: Behavioral: Multiple Channel Exposure Therapy - Veterans
- CPT (Active Comparator): Cognitive Processing Therapy (CPT) is a 12-session cognitive-behavioral treatment for persons with PTSD. It is a gold-standard cognitive behavioral intervention designed to target PTSD symptoms.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Multiple Channel Exposure Therapy - Veterans — MCET-V offers individual therapy that provides psychoeducation about panic attacks and trauma and involves behavioral and cognitive exposure exercises.
  Other Names: MCET-V
  Arms: MCET-V
Behavioral: Cognitive Processing Therapy — CPT offers individual therapy that targets trauma and PTSD symptoms via cognitive restructuring.
  Other Names: CPT
  Arms: CPT

SUMMARY:
To evaluate the feasibility, acceptability and effectiveness of Multiple Channel Exposure Therapy-Veterans (MCET-V) as a treatment for returning service members with comorbid PTSD and panic disorder (PD). This study will examine the effectiveness of MCET-V by comparing it to Cognitive Processing Therapy, a standard PTSD treatment.

DETAILED DESCRIPTION:
With the increasing number of Operations Iraqi Freedom and Enduring Freedom (OIF/OEF) Veterans returning from war-zone areas, many will experience anxiety disorders such as PTSD and comorbid problems. Currently, about one in every six OIF/OEF Veterans experiences PTSD and co-occurring PD. Although effective treatments exist for treating one or the other, we do not yet have treatments that can simultaneously target PTSD and PD. Thus, recent attention has focused on the development of multi-component treatments that simultaneously address PTSD and PD. This study is the first systematic investigation of a time-limited, multi-component cognitive-behavioral treatment for Veterans with specific comorbid anxiety problems. The purpose of the study is to evaluate the effectiveness of the multi-component cognitive-behavioral treatment in comparison to standard PTSD treatment in military personnel returning from active duty.

ELIGIBILITY:
Inclusion Criteria:

* being a Veteran of any era;
* being enrolled in the TRP at the MEDVAMC, with a current diagnosis of PTSD and PD;
* being stable on psychotropic medication for 4 weeks before study participation; and
* being at least 18 years of age.

Exclusion Criteria:

* active substance dependence, or bipolar or psychotic disorders;
* severe depression and [active suicidal ideation and intent] (based on ADIS-IV & BDI-II);
* cognitive impairment as indicated by the SLUMS; and
* Veterans currently receiving psychosocial treatment specifically targeting PTSD or panic symptoms.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Teng, PhD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 93 participants were recruited for the study. Of these participants, 68 met study inclusion criteria and were included in data analyses.
Groups:
- Multiple Channel Exposure Therapy (MCET-V): MCET-V is a 12-session cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks. It is an integrated treatment designed to target panic and PTSD symptoms simultaneously.
- Cognitive Processing Therapy (CPT): CPT is a 12-session cognitive-behavioral treatment for persons with PTSD. It is a gold-standard cognitive behavioral intervention designed to target PTSD symptoms.
Period: Baseline Assessment
Arm/Group | Multiple Channel Exposure Therapy (MCET-V) | Cognitive Processing Therapy (CPT)
Started | 36 | 32
Completed | 30 | 26
Not Completed | 6 | 6
Period: Post-Treatment (1 Week)
Arm/Group | Multiple Channel Exposure Therapy (MCET-V) | Cognitive Processing Therapy (CPT)
Started | 30 | 26
Completed | 16 | 15
Not Completed | 14 | 11
Period: Follow-Up (3 Month)
Arm/Group | Multiple Channel Exposure Therapy (MCET-V) | Cognitive Processing Therapy (CPT)
Started | 16 | 15
Completed | 14 | 13
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiple Channel Exposure Therapy (MCET-V) | Cognitive Processing Therapy (CPT) | Total
Number analyzed (Participants) | 36 | 32 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 29 | 62
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.61 (13.70) | 41.56 (13.26) | 42.12 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 29 | 25 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 12 | 29
  African American | 10 | 13 | 23
  Latino | 7 | 6 | 13
  Asian | 0 | 0 | 0
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms (CAPS) Between MCET-V and CPT Groups
Description: The CAPS is a clinician-administered assessment of the presence and severity of PTSD symptoms. Scores range from 0 - 136, with higher scores indicating greater symptom severity.
Time Frame: Baseline, 1-week post-treatment and 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Multiple Channel Exposure Therapy (MCET-V) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 36 | 32
units on a scale
  Pre-Treatment | 81.8 (21) | 80.5 (19.9)
  Post-Treatment (1 week) | 67.8 (24.2) | 68.1 (26.4)
  Follow-Up (3 months) | 66.6 (20.4) | 66.2 (28.0)
Statistical Analysis 1: Comparison: Multiple Channel Exposure Therapy (MCET-V) vs Cognitive Processing Therapy (CPT); Test type: Equivalence — To test if MCET is equivalent to CPT in decreasing PTSD symptoms, we test the equivalence of the proportion of patients whose CAPS scores decrease by 10 from baseline, by testing whether the difference in proportions between the 2 interventions ≤ to the equivalence margin δb of .20. Results are reported based on 3-month follow-up data; p = 0.30, Fisher Exact — The threshold for statistical significance is p <.05 and is not adjusted for multiple comparisons

2. Primary Outcome: Change in PDSS Scores Over Time for MCET-V and CPT Groups
Description: The Panic Disorder Severity Scale (PDSS) is a clinician-rated assessment of the presence and severity of panic symptoms. Scores range from 0 - 28, with higher scores indicating greater symptom severity.
Time Frame: Baseline, 1-week post, and 3-month follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Multiple Channel Exposure Therapy -Veterans (MCET-V): Multiple Channel Exposure Therapy -Veterans (MCET-V) is a 12-session cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks. It is an integrated treatment designed to target panic and PTSD symptoms simultaneously.
- Cognitive Processing Therapy (CPT): Cognitive Processing Therapy (CPT) is a 12-session cognitive-behavioral treatment for persons with PTSD. It is a gold-standard cognitive behavioral intervention designed to target PTSD symptoms.
Arm/Group | Multiple Channel Exposure Therapy -Veterans (MCET-V) | Cognitive Processing Therapy (CPT)
Number analyzed (Participants) | 36 | 32
units on a scale
  Baseline | 18.5 (3.84) | 16.28 (4.57)
  1-week post | 12.81 (6.33) | 10.20 (5.75)
  3-month follow up | 10.93 (7.53) | 10.62 (6.51)
Statistical Analysis 1: Comparison: Multiple Channel Exposure Therapy -Veterans (MCET-V) vs Cognitive Processing Therapy (CPT); Longitudinal analysis of PDSS scores; Test type: Other; p = 0.68, Mixed Models Analysis — The threshold for statistical significance is p <.05 and is not adjusted for multiple comparisons; Degrees of freedom: 2, 54

ADVERSE EVENTS:
Groups:
- Multiple Channel Exposure Therapy -Veterans (MCET-V): MCET-V is a cognitive-behavioral treatment for persons with comorbid PTSD and panic attacks
  Multiple Channel Exposure Therapy-Veterans: Individual therapy design completed twice a week over a 6-week period. The treatment will include psychoeducation about panic attacks and trauma and behavioral and cognitive exposure exercises.
- Cognitive Processing Therapy (CPT): CPT is a cognitive-behavioral treatment for persons with PTSD
  Cognitive-Processing Therapy: Participants will be randomly assigned to receive either MCET-V or cognitive processing therapy (CPT), a standard PTSD treatment. Patients in both the MCET-V and CPT conditions will receive 12, 90-minute sessions of individual therapy twice a week over a 6-week period.
Arm/Group | Multiple Channel Exposure Therapy -Veterans (MCET-V) | Cognitive Processing Therapy (CPT)
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 0/36 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes